CLINICAL TRIAL: NCT05977751
Title: FINALE: Prospective Multi-Center Trial for FemBloc INtratubal Occlusion for TranscervicAL PErmanent Birth Control
Brief Title: Prospective Multi-Center Trial for FemBloc Permanent Birth Control
Acronym: FINALE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Femasys Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CP-100-009
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Contraception
Keywords: Permanent Birth Control; Permanent Contraception; Permanent Sterilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FemBloc (Experimental): Investigational device and procedure
  Interventions: Device: FemBloc

INTERVENTIONS:
Device: FemBloc — Treatment for women who desire non-surgical permanent birth control by occlusion of the fallopian tubes.

SUMMARY:
Prospective, multi-center, international, unblinded, single-arm trial of subjects undergoing FemBloc followed by ultrasound confirmation test.

DETAILED DESCRIPTION:
Prospective, multi-center, international, unblinded, single-arm trial of subjects undergoing FemBloc followed by ultrasound confirmation test.

ELIGIBILITY:
Inclusion Criteria:

* Female, 21 - 50 years of age desiring permanent birth control.
* Sexually active with male partner.
* Regular menstrual cycle for last 3 months or on hormonal contraceptives.

Exclusion Criteria:

* Uncertainty about the desire to end fertility.
* Known or suspected pregnancy.
* Prior tubal surgery, including sterilization attempt.
* Presence, suspicion, or previous history of gynecologic malignancy.
* Scheduled to undergo concomitant intrauterine procedures (i.e. endometrial ablation) at the time of either FemBloc Treatment or prior to final confirmation test.
* Abnormal uterine bleeding requiring evaluation or treatment.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 573 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Rate | one (1) year
  Number of subjects who were told to rely on FemBloc for birth control and became pregnant through one (1) year.

SECONDARY OUTCOMES:
Reliance Rate | ninety (90) days post treatment
  Number of subjects who were told to rely on FemBloc.
Long term Pregnancy Rate | Five (5) years
  Number of subjects who were told to rely on FemBloc for birth control that became pregnant after one (1) year through 2-, 3-, 4-, and 5-years.

CONTACTS AND LOCATIONS:
Overall Officials: Study Sponsor, Study Director — Medical Affairs and Clinical Development
Locations (6):
- United States (6):
  - Stanford University, Palo Alto, California
  - University of California Davis, Sacramento, California
  - Midtown OB GYN North, Columbus, Georgia
  - Maimonides Medical Center, Brooklyn, New York
  - Seven Hills Women's Health Centers, Cincinnati, Ohio
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: FemBloc Clinical Study Website — http://www.fembloc.com/